CLINICAL TRIAL: NCT01819298
Title: The Influence on Airway Bacteria Colonization in Chronic Obstructive Pulmonary Disease by the Combination of Inhaled Corticosteroid and Long-acting β2 Agonist
Brief Title: Bacterial Colonization in COPD in View of CAT Under ICS+LABA Therapy
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ping-Huai Wang, Doctor, Far Eastern Memorial Hospital
Other Study IDs: FEMH - 2011 - C25
Record Dates: First submitted 2013-03-18; First posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Bacterial Infections; Chronic Obstructive Pulmonary Disease; Self-Assessment
MeSH Terms: conditions — Bacterial Infections; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- bacteria colonization in CAT less 20: the incidence of sputum potential pathogenic microoragnism in patients with CAT scores less than 20
- the PPM in change of CAT >2: the change of potential pathogenic microorganism in CAT difference more than 2 while follow-up
- the change of CAT<=2: the change of potential pathogenic microorganism in CAT difference less than or equal to 2 while follow-up
- PPM in CAT>=20: the incidence of sputum potential pathogenic microoragnism in patients with CAT scores more than or equal to 20

SUMMARY:
Patients with COPD (chronic obstructive pulmonary disease) suffer from episodes of acute exacerbations leading to additional morbidity and mortality, and also a further decline in lung function. It has been well-established that bacterial colonization is prevalent in COPD, especially in moderate to severe COPD, and airway bacterial colonization is known to play an important role in the development of pneumonia and exacerbations. On the other way, inhaled corticosteroid (ICS) and long acting β2 agonist (LABA) were recommended in the treatment of moderate to severe COPD. Though there were some evidences that ICS had some protective effects on airway mucosa against bacteria invasion, the locally immunosuppressive effects of ICS is still a concern. Indeed, the incidence of pneumonia was higher than the control group, not only in the Towards a Revolution in COPD Health (TORCH) study but also in various studies and meta-analyses.We hypothesized that airway bacteria colonization is associated with disease severity, and that disease status can be identified by CAT (COPD assessment test)scores and changes of CAT scores. We therefore conducted this prospective, observational study in which CAT scores and sputum cultures were assessed in moderate to severe COPD patients with the combination therapy of ICS and LABA every three months during the study period. The primary end-point is the condition of potential pathogenic microorganisms (PPM) colonization in view of CAT scores. The second end-point was the changes of PPM colonization in association with CAT changes during follow-up. By the mean of CAT follow-up, it could possibly provide a surrogate about the risk of exacerbation and pneumonia under the combination therapy of ICS and LABA.

ELIGIBILITY:
Inclusion Criteria:

* spirometry showed obstructive ventilatory defect (a ratio of forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) of less than 0.7) and FEV1 less than 80% of predicted value and patients receiving the combination therapy of ICS and LABA

Exclusion Criteria:

* (1) use of antibiotics or corticosteroids within eight weeks before study entry; (2) pneumoconiosis; (3) apparent inactive tuberculosis fibrosis (fibrosis involved in more than one third of one lung field as determined by chest radiography); and (4) asthma and atopic history.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD under ICS+LABA combination therapy and FEV1<80% and FEV1/FVC<70%
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
potential pathogenic microorganisms colonization in view of CAT scores | one year
  Sputum bacterial cultures after sputum induction,and CAT at the start of the study and every three months until the end of the study period

SECONDARY OUTCOMES:
the changes of PPM colonization in association with CAT changes during follow-up. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ping-huai Wang, M.D, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan